CLINICAL TRIAL: NCT06205017
Title: Use of New Food Products (Food for Special Medical Purposes) in the Period Post-bariatric Surgery Weaning to Increase Patient Compliance Diet and Avoid Nutritional Deficiencies.
Brief Title: Post-bariatric Surgery Weaning With Food for Special Medical Purposes to Increase Patient Compliance.
Acronym: AFMS_FOOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AFMS_FOOD (L4190)
Record Dates: First submitted 2023-12-18; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Bariatric Surgery
MeSH Terms: interventions — Food

STUDY DESIGN:
Intervention Model Description: The sample size was calculated in order to identify differences significant in the increase of liking in the study group compared with the control. According to the PI's experience, the frequency of liking in the group control is 5% and this is expected to increase to 70% in the study group.
  Considering using a Fisher's exact test with alpha level=0.05, to obtain a power of 95%, 14 patients per group are needed. This number is increased by 10% in case of possible dropouts, for a total of 16 subjects per group and 32 total.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (AFSM) (Experimental): 16 subjects (Group A: intervention group) will take AFSMs in the immediate postoperative period (Appendix A). A weaning period with AFSM nutritional protocol of 4 weeks is planned, the weaning will cover the entire observation period T0 → T1.
  Interventions: Dietary Supplement: Foods for Special Medical Purposes
- Group B (protocol in use with homogenized) (No Intervention): 16 subjects (Group B: control group) will follow the standard weaning protocol i.e. with homogenized food (Appendix B). A weaning period with nutritional protocol, as per clinical protocol, of 4 weeks is planned, weaning will cover the entire observation period T0 → T1.

INTERVENTIONS:
Dietary Supplement: Foods for Special Medical Purposes — In order to facilitate patient weaning and to improve the enjoyment of foods used in this semi-liquid phase, our Center intends to test "Foods for Special Medical Purposes" (AFMS) to ensure better nutritional intake, including vitamin D3 and calcium, good palatability, and thus better adherence to the recommended nutritional indications in the immediate postoperative period than the homogenized foods used in the standard diet.
  Arms: Group A (AFSM)

SUMMARY:
Due to the reduced volume and postoperative gastric edema, ingestion of solid foods in the first few days after surgery is very difficult or impossible; following bariatric surgery there are anatomical changes in the vagus that may contribute to the alteration of taste perception. In order to facilitate patient weaning and improve the liking of the foods used in this semi-liquid phase, our Center intends to test some "Foods for Special Medical Purposes" (AFMS), in order to ensure a better intake of nutrition, including in terms of vitamin D3 and calcium, good palatability and thus a better adherence to the recommended nutritional indications in the immediate postoperative period than the homogenized foods used in the standard diet.

DETAILED DESCRIPTION:
Primary goal: Patient compliance throughout the weaning period (4 weeks postintervention), assessed through product liking measurable by Sensory Questionnaire.

Secondary objective:

* Patient compliance throughout the weaning period (4 weeks postintervention), assessed through product liking measurable with test comparative
* Taste perception, liking, palatability and food preferences among the different products (Special Medical Purpose Foods-AFMS vs homogenized foods) and between pre and post bariatric surgery.
* Nutritional efficacy (assessment of blood levels of micronutrients such as. iron, ferritin, transferrin , calcium, vit D3, folic ac, vit B12 and of macronutrients such as total protein and protein electrophoresis; bioimpedance analysis for body composition assessment).

  32 subjects with severe or morbid obesity ( BMI ≥ 35 kg/m2 in the presence of comorbidities and BMI ≥ 40 kg/m2 , respectively), male and female, candidates for bariatric surgery (Sleeve Gastrectomy and Roux-en-Y Gastric Bypass).

Two timepoints: T0 (pre-rev) and T1 (follow-up 1 month +/-7 days). Planned assessments at T0 and T1.

* Administration of the sensory questionnaire.
* Comparative test
* Hematochemical tests: iron, ferritin, transferrin, , vit D3, ac. Folic, vit B12 and macronutrients such as total protein + general hematochemicals (complete blood count complete, protein electrophoresis, AST, ALT, gamma GT, creatininemia, azotemia, col tot, HDL, LDL, triglycerides, blood glucose).
* Analysis of taste perception and variation by Taste Strips.
* Bioimpedance analysis (BIA)
* Anthropometric evaluations

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤ of 60
* Subjects with severe or morbid obesity (BMI ≥ 35 kg/m2 in the presence of comorbidities and BMI ≥ 40 kg/m2)
* Absence of diagnosis of primary obesity
* Absence of medical/psychiatric contraindications
* Signature of informed consent for the study
* Patients who are candidates by clinical practice for bariatric surgery (Sleeve Gastrectomy and Roux-en-Y Gastric Bypass).

Exclusion Criteria:

* Presence of chronic diseases of the digestive system, such as chronic diseases intestinal, malabsorption syndrome, diverticulosis of the colon
* Current pregnancy (verified by self-declaration) and/or lactation
* Subjects with endocrine disorders (e.g., Cushing's m., thyroid disease uncontrolled)
* Presence of known renal insufficiency or creatinine levels greater than 1.8 mg/dl and eGFR < 60 ml/min
* Presence of malignant pathology
* Alcohol or drug abuse
* Severe psychological/psychiatric disorders
* Difficulty adhering to the protocol due to language barriers or other reasons.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-01-09 (Estimated); Primary Completion 2024-07-09 (Estimated); Study Completion 2024-08-09 (Estimated)

PRIMARY OUTCOMES:
Patient compliance throughout the weaning period | 1 month
  Patient compliance throughout the weaning period (4 weeks post-intervention), assessed through satisfaction with the products measurable with a questionnaire sensory.

IPD SHARING:
Plan to Share IPD: No